CLINICAL TRIAL: NCT01642017
Title: Phase I Clinical and Pharmacokinetic Study of Pazopanib in a Population of Frail Elderly Patients According SIOG Criteria
Acronym: VOTRAGE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11GENE06
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Cancer (Different Solid Tumour Types)
Keywords: Phase I, Pazopanib, Frail elderly patients, Pharmacokinetics
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib (Experimental): Pazopanib : 3 dose levels are defined : 400, 600 and 800 mg per day.
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Pazopanib will be administered orally at the starting dose of 400 mg/day in 28-days cycles ; barring limiting toxicities the dose of pazopanib will escalate in several steps (a maximum of 3 dose levels are defined : 400, 600 and 800 mg/day). The pazopanib will be administered at the same dosa until disease progression.

SUMMARY:
This is an open-label, multicenter, non-randomized, phase 1 dose escalation clinical trial to determine the MTD (Maximal Tolerated Dose) of Pazopanib in a population of frail elderly patients, selected according to the International Society of Geriatric Oncology (SIOG)classification (Group 2).

It is expected that a total number of 30 patients maximum will be enrolled in the study on 30 months : 18 months accrual - 12 months follow up.

Eligible patients will be enrolled into a standard 3+3 design with a starting dose of Pazopanib administered orally at 400 mg per day, in 28-day cycles. Then, further dose levels will be explored.

Toxicity of the schedule will be assessed during the first cycle. Patients will receive study medication until disease progression. After treatment discontinuation, patients will be followed during one year.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow up.
2. Age ≥ to 75 years old
3. Patient with metastatic cancer among renal cell carcinoma, non small cell lung cancer, pancreatic neuroendocrine cancer, sarcoma , ovarian cancer , thyroid cancer, bladder cancer or breast cancers, who cannot receive any treatment with curative intent.
4. WHO PS ≤ 2,
5. Life expectancy ≥ 3 months,
6. Group 2 (vulnerable) according to SIOG classification,
7. Adequate organ system function as defined in provided Table

Exclusion Criteria:

1. Patient with a history of a prior malignancy with the exception of cervical intraepithelial neoplasia; basal cell carcinoma of the skin; adequately treated localized prostate carcinoma with PSA <1.0; or who has undergone potentially curative therapy with no evidence of that disease for five years, and who is deemed at low risk for recurrence by his/her treating physician,
2. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug.
3. Criteria of group 3 according to SIOG classification,
4. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

   •Active peptic ulcer disease

   •Known intraluminal metastatic lesion/s with risk of bleeding

   •Inflammatory bowel disease (e.g. ulcerative colitis, crohn's disease), or other gastrointestinal conditions with increased risk of perforation

   •History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
5. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

   •Malabsorption syndrome

   •Major resection of the stomach or small bowel.
6. Presence of uncontrolled infection.
7. Corrected QT interval (QTc) > 480 msecs using Bazett's formula
8. Anti-coagulants treatment (preventive or curative)
9. History of any one or more of the following cardiovascular conditions within the past 6 months:

   • Cardiac angioplasty or stenting

   • Myocardial infarction

   • Unstable angina

   • Coronary artery bypass graft surgery
   * Symptomatic peripheral vascular disease
   * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
10. Poorly controlled hypertension
11. History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
12. Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer
13. Evidence of active bleeding or bleeding diathesis.

14 Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels

15. Hemoptysis in excess of 2.5 mL (or one half teaspoon) within 8 weeks of first dose of study drug.

16. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.

17. Unable or unwilling to discontinue use of prohibited medications list in Appendix 7 for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study

18. Treatment with any of the following anti-cancer therapies:

* radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR
* chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib

  19. Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia.

  20. Patient not affiliated with social system in France.

  21. Patient deprived of liberty or under guardianship

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-11-22 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) incidence (according DLT definition) during the first treatment cycle with pazopanib (28 days) | 7.5 years
  The MTD (Maximum Tolerated Dose) is defined as the highest dose level for which 6 patients were treated with a maximum of 1 patient presenting a DLT during the first cycle of treatment

SECONDARY OUTCOMES:
Safety and tolerability assessments using the descriptions and grading scales found in the CTCAE (Common Terminology Criteria for Adverse Events) version 4.0 NCI | 7.5 years
Measure of Pazopanib plasma concentration during treatment period (objective : assessment of pharmacokinetics of Pazopanib in this population) | .8 time points (cycle 1 Day 1), 3 time points (cycle 1 D15) and 1 pre dose time point each day 1 of the following cycles (over a period of 7.5 years for measures in all patients)
  Plasma concentrations of pazopanib will be determined using a validated LC-MS-MS method -
Geriatric criteria measured by comprehensive geriatric assessment which evaluate medical, functional and psychosocial aspects of elderly patients | 7.5 years
  The impact of treatment on the geriatric assessment will be done using :
  * G8 : screening test
  * ADL: Activities Daily Living
  * IADL: Instrumental Activities Daily Living
  * MMSE: Mini-mental State Examination
  * SPPB: Short Physical Performance Battery
  * MNA: Mini-nutritional Assessment
  * CAM: Confusion Assessment Method
  * GDS-15: Geriatric Depression Scale
  * CIRS-G: Cumulative Illness Rating Scale for Geriatrics,
Rate of objective response according to RECIST criteria | 7.5 years
  Tumor assessment will be performed at screening visit, every 2 cycles and at the end of study visit and anytime if clinically indicated

CONTACTS AND LOCATIONS:
Overall Officials: Loïc MOUREY, PhD, Principal Investigator — Institut Claudius Regaud
Locations (4):
- France (4):
  - Hôpital Saint André, Bordeaux
  - Centre François BACLESSE, Caen
  - Centre Léon BERARD, Lyon
  - Institut Claudius REGAUD, Toulouse